CLINICAL TRIAL: NCT01140386
Title: Prevalence and Risk Factors of Venous Thromboembolism in Hospitalized Pediatric Patients
Acronym: pediatric DVT
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Other Study IDs: 30835
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2010-06

CONDITIONS: Venous Thromboembolism; Deep Venous Thrombosis; Pediatrics
Keywords: venous thromboembolism; duplex ultrasound; pediatric population; Vascular lab duplex ultrasound database; Inpatient hospital admission/discharge ICD-9 database; PTSF pediatric trauma database
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hospital pediatric patients 1/1/2000-12/31/2008 documented VTE: Age <18 Hospitalized for greater than or equal to 24 hours VTE documented during hospital admission

SUMMARY:
The issue to be studied is the prevalence of venous thromboembolism (VTE) in hospitalized pediatric patients, and to identify if there are subgroups of patients who may be at higher risk.

There are two hypotheses that will be looked at in this study. The first hypothesis is that individual risk factors for VTE in hospitalized pediatric patients are: age >14, obesity, black race, female sex, presence of a central venous line (CVL), traumatic mechanism of injury, orthopaedic surgery, and use of oral contraceptives.

The second hypothesis is that risk factors have an additive effect such that risk stratification can be developed to identify those patients with the highest risk.

DETAILED DESCRIPTION:
Venous thromboembolism is a well recognized concern in the hospitalized adult population: 11-15% of medically ill adults will have venous thromboembolism (VTE) and 4-5% will develop a proximal DVT in the absence of prophylaxis.6 Furthermore, these diagnosed events are an underestimation of the prevalence of VTE as 80% are clinically silent.6 VTE risk stratification exists for adult populations and prophylaxis against VTE is standard procedure. While VTE occurs less frequently in pediatric populations, the incidence is on a rise. Vu et al report a significant increase in DVT in 2003 compared to 1997 using data from the Health Care Cost and Utilization Project Kids' Inpatient Database. 2 If one were to extrapolate the known adult risk factors for VTE to children, this rise could be attributed to an increase in childhood obesity ,4 an increase in estrogen-based therapy among teenage girls1, or the increase in pediatric trauma.3 However, few studies have been performed to show if these or other identified adult risk factors are indeed pediatric risk factors as well. Due to this lack of knowledge of risk factors for VTE in pediatric populations, there are minimal guidelines for when physicians should provide prophylactic treatment or even have heightened awareness of the possibility of VTE in their pediatric patient. Furthermore, there are scant published guidelines regarding which type of prophylactic treatment is safe and efficacious in the pediatric population, nor are there guidelines regarding the treatment of established VTE. Outcomes of prophylactic treatment will not be able to be evaluated accurately until the measures are undertaken in patients with identified high risk. Identification of high risk groups and subsequent prevention of VTE is important due to the significant morbidity and mortality associated with VTE. Vu et al report a two-fold increase in in-hospital death in pediatric patients with an identified VTE compared to those without one. This risk was independent of other comorbid conditions.2 Morbidity includes pulmonary embolism, recurrent thrombosis, and postphlebitic syndrome (characterized by swelling, pain, skin indurations and pigmentation caused by incompetent venous valves). Due to the younger age of onset, pediatric patients with these morbidities live with the consequences for a much longer period of time; furthermore, they may experience secondary consequence such as limb length discrepancies, etc.

Currently there is a sharp delineation in prophylaxis strategy as defined merely by age. As soon as a patient is 18 he is assessed by risk stratification models and given prophylaxis if he meets these criteria. A patient just one year younger, however, is left unevaluated due to the lack of criteria for VTE risk in pediatric patients. The patient may fit height and weight averages of a full grown adult, and may possess many of the criteria used to assess an adult for VTE risk. He still may not be offered prophylaxis treatment due to his age alone. This assumes age is the best predictive factor of VTE in the younger patient. However, few studies have been done assessing what risk factors truly exist for the pediatric patient, and those that have, suggest that there are other factors that play into the equation, and may even be more important.5 Due to potential complications from both VTE as well as prophylaxis, and the increasing prevalence of VTE in pediatric populations, studies regarding risk factors and safety/efficacy of prophylactic treatment are needed to establish guidelines of care.

ELIGIBILITY:
Inclusion Criteria:

* Age <18
* Hospitalized for greater than or equal to 24 hours
* VTE documented during hospital admission

Exclusion Criteria:

* Age >18

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients aged <18 years old, who were hospitalized at MSHMC from January 1, 2000 -December 31, 2008 with documented VTE in one of three databases:
  1. Vascular lab duplex ultrasound database
  2. Inpatient hospital admission/discharge ICD-9 database
  3. PTSF pediatric trauma database
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
documented deep vein thrombosis (DVT) | 1/1/200 - 12/31/2008
  Patients aged <18 years old, who were hospitalized at MSHMC from January 1, 2000 -December 31, 2008 with documented VTE in one of three databases:
  1. Vascular lab duplex ultrasound database
  2. Inpatient hospital admission/discharge ICD-9 database
  3. PTSF pediatric trauma database

REFERENCES:
- [Result] Department of Health and Human Services, Centers for Disease Control and Prevention: http://www.cdc.gov/nchs/data/series/sr_23/sr23_024.pdf 2. L.T. Vu, K.K. Nobuhara, and H. Lee et al., Determination of risk factors for deep venous thrombosis in hospitalized children. Journal of Pediatric Surgery 43 (2008), pp 1095-1099. 3. M.S. Vavilala, A.B. Nathens and G.J. Jurkovich et al., Risk factors for venous thromboembolism in pediatric trauma, J Trauma 52 (2002), pp. 922-927 4. National Health and Nutrition Exam Survey (NHANES); Dept of Health and Human Services, Centers for Disease Control and Prevention: http://www.cdc.gov/nccdphp/dnpa/obesity/childhood/prevalence.htm 5. P.D. Stein, F. Kayali and R.E Olson et al. Incidence of venous thromboembolism in infants and children: Data from the National Hospital Discharge Survey, The Journal of Pediatrics 145 (2004), pp 563-565. 6. R. Pendleton, M. Wheeler, and G. Rodgers. Venous Thromboembolism Prevention in the Acutely Ill Medical Patient: A Review of the Literature and Focus on Special Patient Populations, American Journal of Hematology 79 (2005), pp 229-237.